CLINICAL TRIAL: NCT04549649
Title: Royan Institute for Reproductive Biomedicine
Brief Title: The Effect of Dual Trigger for Final Oocyte Maturation on IVF/ICSI Outcomes in Patients With Suboptimal Ovarian Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Research ID (96000024)
Record Dates: First submitted 2020-08-05; First posted 2020-09-16 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Stimulation; Reproductive Techniques, Assisted
Keywords: Poor ovarian response; Dual trigger; GnRH antagonist protocol
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental oocyte triggering approach) (Experimental): 0.2 mg Triptorelin (Decapeptyl; Ferring GmbH) associated with two ampoules of Ovitrelle (Ovitrelle®, 250 μg/0.5 ml, Merck, Serono, Inc) will be administered subcutaneously simultaneously for final oocyte triggering.
  Interventions: Other: Dual triggering
- Group B (Routine oocyte triggering approach) (No Intervention): Two ampoules of Ovitrelle® (Ovitrelle®, 250 μg/0.5 ml, Merck, Serono, Inc) will be injected subcutaneously for final oocyte triggering.

INTERVENTIONS:
Other: Dual triggering — Adding GnRH agonist (0.2 mg Triptorelin (Decapeptyl; Ferring GmbH) to routine oocyte triggering (two ampoules of Ovitrelle®, 250 μg/0.5 ml, Merck, Serono, Inc) is defined as dual triggering.
  Arms: Group A (Experimental oocyte triggering approach)

SUMMARY:
Recently, in patients with a suboptimal ovarian response, a study of the role of adding a single dose of GnRH agonist to a standard dose of hCG to initiate final oocyte maturation has also been studied. Griffin et al. (2014) reported that in patients who had more than 25% immature oocytes in their previous IVF cycle, the use of dual stimulation could increase the number of mature oocytes. Since studies in this field are limited, the researchers decided to design a clinical trial to investigate the effect of adding a GnRH agonist to a standard dose of hCG to initiate final oocyte maturation in patients with a sub-optimal ovarian response.

DETAILED DESCRIPTION:
Ovulation stimulation will be performed in all patients with the Standard GnRH antagonist Protocol with E2 priming, with the antagonist protocol administered in all patients from the 20th cycle until the start of the next menstrual cycle with 4 mg of estradiol daily. Blood sampling (FSH, LH, and estradiol levels) will be performed on the second day of the menstrual cycle, just before gonadotropin stimulation. Ovarian stimulation will start from the second or third day of menstruation with a maximum dose of 225 units of rFSH (Gonal -F: Serono Laboratories Ltd, Geneva, Switzerland), and then if the follicle is observed, start with 13 injections of GnRH antagonist (Cetrotide®, 0.25 mg cetrorelix acetate, Serono, Inc)). From the seventh day of the cycle, the dose of rFSH will be determined according to the rate of ovarian response by vaginal ultrasonography two days in advance. If you see at least 2 follicles 18 mm in size or more, the antagonist will be injected. GnRH and gonadotropins (Gonal-F) will stop and (oocyte triggering) will be the final stimulation of oocyte maturation, at this time, the block randomization method will be designed to randomize allocation of patients into groups with blocks of size 4. Recently, in patients with a suboptimal ovarian response, a study of the role of adding a single dose of GnRH agonist to a standard dose of hCG to initiate final oocyte maturation has also been studied. Griffin et al. (2014) reported that in patients who had more than 25% immature oocytes in their previous IVF cycle, the use of dual stimulation could increase the number of mature oocytes. Since studies in this field are limited, the researchers decided to design a clinical trial to investigate the effect of adding a GnRH agonist to a standard dose of hCG to initiate final oocyte maturation in patients with a suboptimal ovarian response.

Controlled Ovulation stimulation (COS) will be performed in all patients with the Standard GnRH antagonist Protocol with E2 priming, with the antagonist protocol administered in all patients from the 20th cycle until the start of the next menstrual cycle with 4 mg of estradiol daily. Blood sampling (FSH, LH, and estradiol levels) will be performed on the second day of the menstrual cycle, just before gonadotropin stimulation. Ovarian stimulation will start from the second or third day of menstruation with a maximum dose of 225 units of rFSH (Gonal -F: Serono Laboratories Ltd, Geneva, Switzerland), and then if the follicle is observed, start with 13 injections of GnRH antagonist (Cetrotide®, 0.25 mg cetrorelix acetate, Serono, Inc)). From the seventh day of the cycle, the dose of rFSH will be determined according to the rate of ovarian response by vaginal ultrasonography two days in advance. If you see at least 2 follicles 18 mm in size or more, the antagonist will be injected. GnRH and gonadotropins (Gonal-F) will stop and (oocyte triggering) will be the final stimulation of oocyte maturation, at this time, the block randomization method will be designed to randomize allocation of patients into groups with blocks of size 4. The required number of blocks will be randomly selected according to sample size.

The final ovarian stimulation (oocyte triggering) will be performed in groups A and B as follows:

Group A (Experimental): 0.2 mg Triptorelin (Decapeptyl; Ferring GmbH) associated with two ampoules of Ovitrelle (Ovitrelle®, 250 μg/0.5 ml, Merck, Serono, Inc) will be administered subcutaneously simultaneously.

Group B (Control): Two ampoules of Ovitrelle® (Ovitrelle®, 250 μg/0.5 ml, Merck, Serono, Inc) will be injected subcutaneously.

The COS cycles with less than two follicles will be cancelled s. Ovum pick up is performed 32-34 hours after oocyte triggering, and subsequently intracytoplasmic sperm injection (ICSI) /in-vitro fertilization (IVF) will be done for all the patients.

The main outcome measures are the number of dominant follicles (≥13 mm) on the day of hCG trigger and the number of mature (MII) oocytes collected after conventional versus delayed-start ovarian stimulation protocol. Secondary outcome measures are including total number of oocytes retrieved, oocyte maturity rate (number of MII oocytes/total number of oocytes), oocyte yield (total number of oocytes retrieved/ antral follicle count [AFC]), mature oocyte yield (number of mature oocytes retrieved/AFC), total dosage of gonadotropin (recombinant FSH and/or highly purified hMG) needed, number of days needed for ovarian stimulation, quality of obtained embryos, fertilization rate (the proportion of total number of two-pronuclear [2PN] stage zygotes /per total injected MII oocytes), implantation rate (total number of observed gestational sac/ number of transferred embryos) and clinical pregnancy rate (presence of fetal heart beat by transvaginal ultrasound per embryo transfer).

ELIGIBILITY:
Inclusion Criteria:

Patients with poor ovarian response (POR) diagnosis according to the POSEIDON stratification system (as POSEIDON group 1) with following criteria :

* Women' age under 35 years;
* Previous unexpected poor or suboptimal ovarian response after using conventional protocols (subgroup 1a: < 4 oocytes ) and (subgroup 1b: 4-9 oocytes retrieved)
* Adequate ovarian reserve (antral follicle count ≥5 on menstrual cycle day 2-3; and basal serum AMH ≥ 1.2 ng/ml)

Exclusion Criteria:

* Ovarian failure including basal FSH above 20 IU/l or no antral follicle by ultrasound examination;
* Endometriosis grade 3 or higher;
* Severe male infertility (surgical sperm extraction: TESE, PESA)
* Body mass index >30 kg/ m2
* History of uterine surgery as well as sub-mucosal and intramural fibroids greater than 5 cm or uterine polyps
* Treatment cycles with pre-implantation genetic diagnosis, blastocyst and donation embryo transfer indications
* Cigarette and drug addiction

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Total number of retrieved oocytes | Day of oocyte pick-up (32-34 hours after hCG administration)
  In one hour after ovum pick-up, outcome measurement will be possible.
Total number of mature or metaphase II (MII) oocytes | Day of oocyte pick-up ( 32-34 hours after hCG administration )
  In one hour after ovum pick-up, counting the total number of MII oocytes will be possible.
Oocyte recovery ratio | 32-34 hours after oocyte triggering
  Ratio of the total number of follicles above 18 mm to the total number of retrieved oocytes

SECONDARY OUTCOMES:
Fertilization rate | Day 1 post oocyte retrieval
  The number of 2 pronucleus (2pn) oocytes per number of injected and/or inseminated MII oocytes
Quality of obtained embryos: grade | 3 days after in vitro fertilization/ intracytoplasmic sperm injection (IVF/ICSI) procedure
  The quality of embryos was graded from 1 to 3 under inverted microscope 3 days after IVF/ICSI procedure. Embryos with even-sized blastomers and/or ≤10% fragments were classified as Grade 1 (Excellent or good quality). Grade 2 embryos (moderate or fair quality) had blastomeres with slightly-moderate size differences and/or 10- 20% fragments. Grade 3 embryos (poor quality) had markedly different-sized blastomers and/or >20% fragments.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Hafezi, M.D., Principal Investigator — Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
The principle investigator of study can share IPD after finishing the study and publishing the results.
Supporting Information: Study Protocol, SAP
Time Frame: After finishing the study and publishing the results.
Access Criteria: Contact the principal investigator by Email.

REFERENCES:
- [Derived] Hafezi M, Arabipoor A, Zareei M, Vesali S, Mostafaei P, Zameni N. The Effect of Dual Trigger on In Vitro Fertilization/Intracytoplasmic Sperm Injection Outcomes in Patients with Suboptimal Ovarian Response (POSEIDON Classification Group I): A Randomized Clinical Trial. Int J Fertil Steril. 2025 May 14;19(3):251-258. doi: 10.22074/ijfs.2025.2027114.1669. PMID 40590283